CLINICAL TRIAL: NCT00933374
Title: A Single Arm, Multi-center Phase II Trial to Evaluate Paclitaxel Plus RAD001 in Urothelial Carcinoma After Failure of Prior Platin-based Chemotherapy
Brief Title: Trial to Evaluate Paclitaxel Plus RAD001 in Urothelial Carcinoma
Acronym: RAD001
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: delayed recruitment
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001L DE 17T
Record Dates: First submitted 2009-07-03; First posted 2009-07-07 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; RAD001; Paclitaxel
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Paclitaxel; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel and RAD001 (Experimental): 175 mg /m3 paclitaxel every 3 weeks and 10 mg RAD001 once daily starting at day 1 of a 21 days treatment cycle
  Interventions: Drug: paclitaxel; Drug: RAD001

INTERVENTIONS:
Drug: paclitaxel — Paclitaxel (175 mg/m3)will be administered as a 3 hour continuous IV infusion after standard premedication every 3 weeks
  Other Names: Taxol
Drug: RAD001 — 10 mg RAD001 once daily starting at day 1 of a 21 days treatment cycle
  Other Names: Certican, Everolimus

SUMMARY:
This is a single arm open- label phase II- trial evaluating safety and efficacy of paclitaxel and RAD001 in patients with metastatic urothelial bladder cancer who failed prior platin-based systemic therapy.

DETAILED DESCRIPTION:
The screening phase for checking eligibility and evaluation of the patient prior start of study treatment will last up to 21 days.Tumor histology must be predominant urothelial carcinoma and confirmed histological or cytological.Patients who meet the inclusion criteria will be treated with paclitaxel 175 mg/m2 every 3 weeks and RAD001 10 mg once daily. Each cycle will use the combination of paclitaxel 175 mg/m2 3-weekly with RAD001 10 mg daily starting at day 1 of a 21 days treatment cycle. Additional visits after day 1 are performed at day 8 and day 15 of each cycle Assessment of safety and toxicity will be performed at every visit.

Patients will be treated until no signs of clinical or radiological progression are evident and the study treatment is well tolerated for a maximum of 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven carcinoma of the urinary tract including urinary bladder, ureter, renal pelvis and lower urinary tract. Urothelial carcinoma should be the predominant histology
* Confirmation of locally relapsed or metastatic disease by imaging. Measurable disease according to RECIST- guidelines with ≥1 measurable lesion has to be evident.
* If bone is the only metastatic site a quantification of the target lesion(s) using MRI is mandatory.
* Failure of prior platin- based chemotherapy
* Patients may have shown progressive disease within the first 3 months of platin-based chemotherapy (primary failure) or progression within 3 months after the end of platin-based chemotherapy (early relapse)-Prior therapy with ≤ 4 chemotherapeutic drugs
* Patients with tumor relapse within 3 months after cystectomy in the neoadjuvant or adjuvant setting are not eligible.
* ECOG performance status 0-2
* Adequate haematological, liver and renal functions.

  * Neutrophil count > 1500/mm3, haemoglobin > 9 g/dl, platelets ≥ 100.000/ mm3
  * Serum bilirubin ≤ 1.5 x ULN, ALT and AST ≤ 2.5x ULN. Patients with known liver metastases who have an AST and ALT ≤ 5x ULN.
  * serum creatinine ≤ 2 x ULN.
* Women of childbearing potential must have a negative serum or urine pregnancy test within 14 days prior to the first dose of study drug. Female subjects of childbearing potential must be using two acceptable methods of contraception, from the time of screening and for the duration of the study, through study completion and for 3 months following study completion
* Age > 18 years.
* Able to communicate well with the investigator, to understand and comply with the requirements of the study. Understand and sign the written informed consent.
* Patients must give written informed consent
* No concurrent treatment with other experimental drugs or anti-cancer drugs
* Another distinguishable malignancy will be permitted

Exclusion Criteria:

* chemotherapy, radiation therapy or any other anticancer therapy within 4 weeks of the first dose of study drug.
* Participation in any clinical investigation within 4 weeks prior to initial dosing.
* known hypersensitivity to RAD001 or other rapamycin analogs and paclitaxel or other taxanes, or to its excipients.
* previously received RAD001, other mTOR inhibitors or taxanes or epothilones
* known metastasis of central nervous system.
* symptomatic pleural effusions or symptomatic ascites.
* wide field radiation therapy to up to ≥ 25% of the bone marrow within 4 weeks prior therapy.
* intravenous radionuclide therapy, e.g. phosphorus (32P), strontium (89SrCl), rhenium (186Re)or samarium (153Sm).
* Patients who have undergone major surgery within 4 weeks prior to starting study drug,open biopsy, or significant traumatic injury, or who have not recovered from the side effects of any of the above.
* Chronic systemic treatment with corticosteroids corresponding to a prednisone equivalent of > 10 mg daily. Patients receiving corticosteroids must be on a stable dose for ≥ 4 weeks prior to the first dose of RAD001. Topical or inhaled corticosteroids are permitted.
* Concomitant medication with strong CYP3A4- inhibitors or CYP3A4- inducers.
* active bleeding diathesis.
* Neuropathy > grade 1.
* any severe and/or uncontrolled medical conditions(unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤ 6 months, serious uncontrolled cardiac arrhythmia, uncontrolled hyperlipidemia, active or uncontrolled severe infection,cirrhosis,chronic or persistent active hepatitis)
* severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or O2 saturation ≤ 88% at rest on room air
* Uncontrolled diabetes
* Hepatic impairment with a Child-Pugh score >9

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-07; Primary Completion 2013-01 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Response rate | 3 years

SECONDARY OUTCOMES:
Duration of response | from first determination of response until progression
Progression free survival | 3 years
overall survival | 3 years
safety profile of combination RAD001 and paclitaxel | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Peter Albers, Professor, Principal Investigator — Heinrich-Heine-University, Department of Urology
Locations (6):
- Germany (6):
  - Klinik für Urologie, Klinikum rechts der Isar der TU München, München, Bavaria
  - Universitätsklinik Hamburg, Medizinische Klinik und Poliklinik Onkologie - Hämatologie, Hamburg, Hamburg
  - Heinrich-Heine-University of Duesseldorf, Department of Urology, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinik Essen, Klinik für Urologie, Essen, North Rhine-Westphalia
  - Klinik für Urologie, Universitätsklinikum Muenster, Münster, North Rhine-Westphalia
  - Klinik für Urologie und Kinderurologie, Universitätsklinikum des Saarlandes, Homburg, Saarland